CLINICAL TRIAL: NCT05896774
Title: AN OPEN-LABEL, PHASE 1 STUDY EVALUATING THE PHARMACOKINETICS, SAFETY AND ANTI-TUMOR ACTIVITY OF PF-07901801 (TTI-622) MONOTHERAPY IN CHINESE PARTICIPANTS WITH ADVANCED HEMATOLOGIC MALIGNANCIES
Brief Title: A Study to Learn About the Study Medicine (Maplirpacept) in People With Advanced Non-Hodgkin Lymphoma or Multiple Myeloma in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C4971010
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Non-Hodgkin Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maplirpacept (PF-07901801) (Experimental): single arm study
  Interventions: Drug: Maplirpacept

INTERVENTIONS:
Drug: Maplirpacept — Study drug will be administered intravenously with adjustment for body weight weekly over 28-day cycles.
  Other Names: PF-07901801; TTI-622

SUMMARY:
The purpose of this study is to learn about the safety and what the body does to the medicine (Maplirpacept) when taken for the treatment of non-Hodgkin lymphoma or multiple myeloma.

Non-Hodgkin lymphoma is any of a large group of cancers of lymphocytes (white blood cells). Multiple myeloma is a type of cancer that begins in plasma cells (white blood cells that produce antibodies).

This study is seeking participants who:

* have non-Hodgkin lymphoma or multiple myeloma.
* have worsened with (or lack of improvement to) a standard treatment taken before.
* have relatively normal functioning organs.

All participants in this study will receive Maplirpacept as an intravenous (IV) infusion (given directly into a vein) at the study clinic every week.

Participants will continue to receive Maplirpacept until:

* the cancer worsens.
* some serious side effects show up.
* the participants do not wish to take the study medicine any more.

The experiences of the people receiving the study medicine will be collected. This will help to understand if the study medicine Maplirpacept, is safe and can be given to Chinese people.

DETAILED DESCRIPTION:
The study is composed of 2 parts. In Part A, approximately 3-6 participants are expected to be enrolled to confirm the tolerability in Chinese participants. If deemed safe, the enrollment of Part B will proceed to include a total of approximately 9 participants in the study to continue to evaluate the pharmacokinetics, safety and preliminary efficacy of single agent PF-07901801 (Maplirpacept).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed relapsed/refractory non-Hodgkin lymphoma without other effective therapeutic option. Or relapsed/refractory multiple myeloma exposed to therapies including PI, IMiD and anti-CD38 antibody.
* With measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
* Adequate organ functions (including hematologic status, coagulation, hepatic, and renal)

Key Exclusion Criteria:

* Active plasma cell leukemia, or POEMS syndrome.
* Known, current central nervous system disease involvement.
* Significant cardiovascular disease.
* Chronic use of systemic corticosteroids of more than 20 mg/day of prednisone or equivalent.
* Radiation therapy within 14 days of study treatment administration.
* Hematopoietic stem cell transplant within 90 days before the planned start of study treatment or participants with active GVHD disease.
* Use of any anticancer drug within 14 days before planned start of study treatment.
* Prior anti-CD47 or anti-SIRP alpha therapy.
* Participation in other studies involving investigational drug(s) or vaccines within 4 weeks from the last dose
* Known active, uncontrolled bacterial, fungal, or viral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose-Limiting Toxicity (DLT) | Cycle 1：up to 21 days
  Part A only. To characterize the dose limiting toxicities (DLTs) of Maplirpacept.
Single-dose Cmax | 0, 1, 2, 4, 24, 72 hours post-dose up to Day 8
  Maximum Observed Plasma Concentration
Single-dose AUClast | 0, 1, 2, 4, 24, 72 hours post-dose up to Day 8
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Single-dose AUCtau | 0, 1, 2, 4, 24, 72 hours post-dose up to Day 8
  Area under the concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 1 week.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) by type, frequency, severity (as graded by NCI CTCAE verision 5.0), timing, seriousness and relationship to study treatment | Baseline up to 28 days after the last dose of study drug
  An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Participants with multiple occurrences of an AE within a category were counted once within the category. Relatedness to study drug was assessed by the investigator.
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing | Baseline up to 28 days after the last dose of study drug
  Laboratory parameters included: hematology, blood chemistry and coagulation. Clinical significance of laboratory parameters was determined at the investigator's discretion.
Single-dose Tmax (Time to Reach Maximum Observed Plasma Concentration) | 0, 1, 2, 4, 24, 72 hours post-dose up to Day8
  Pharmacokinetics of Maplirpacept
Multiple-dose Cmax (Maximum Observed Plasma Concentration) | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
Multiple-dose Ctrough (trough concentration) | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
Multiple-dose Cmin (Minimum Observed Plasma Trough Concentration) | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
Multiple-dose Tmax (Time to Reach Maximum Observed Plasma Concentration) | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
Multiple-dose AUClast (Area under the plasma concentration time-curve from zero to the last measured concentration) | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
Multiple-dose AUCtau (Area Under the Curve from Time Zero to end of dosing interval) | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
Multiple-dose Rac (Accumulation Ratio) | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
CL (Systemic Clearance) | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
Vss (Volume of Distribution at Steady State) | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
t½ (Plasma Decay Half-Life) | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
AUCinf (Area Under the Curve From Time Zero to Extrapolated Infinite Time) | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
Incidence and titers of anti-drug antibodies against TTI-622 | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
Incidence and titers of neutralizing antibodies against TTI-622 | Through study completion, up to 18 months
  Pharmacokinetics of Maplirpacept
Objective Response | Baseline to measured progressive disease, up to 18 months
  To assess the preliminary antitumor activity of Maplirpacept
Time to Tumor Response (TTR) | Baseline to measured progressive disease, up to 18 months
  To assess the preliminary antitumor activity of Maplirpacept
Duration of Response (DOR) | Baseline to measured progressive disease, up to 18 months
  To assess the preliminary antitumor activity of Maplirpacept
Progression-Free Survival (PFS) | Baseline to measured progressive disease, up to 18 months
  To assess the preliminary antitumor activity of Maplirpacept
Minimal Residual Disease (MRD) | Baseline to measured progressive disease, up to 18 months
  To assess the preliminary antitumor activity of Maplirpacept. Multiple myeloma participants achieved complete response will be assessed for MRD status per IMWG MRD criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4971010